CLINICAL TRIAL: NCT06055387
Title: Frailty Assessment and Intervention in Elderly Patients with Gastric Cancer Receiving Gastrectomy and Adjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202101510B0C601
Record Dates: First submitted 2023-08-29; First posted 2023-09-26 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
Keywords: Frailty; Comprehensive Geriatric Assessment (CGA); Outcome; Radical surgery; Adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frail group (Experimental): All patients receive a frailty assessment within 7 days before initiating treatment, followed by geriatric intervention. Patients exhibiting impairments in at least two dimensions are considered frail. The frail group will receive management and recommendations based on the specific impairment domain.
  Interventions: Behavioral: Frailty intervention measures
- Non-frail group (No Intervention): All patients receive a frailty assessment within 7 days before initiating treatment, followed by geriatric intervention. Patients exhibiting impairments in at least two dimensions are considered frail. The non-frail group will not receive additional interventions, but the clinical physicians will still provide appropriate treatment based on the patient's condition.

INTERVENTIONS:
Behavioral: Frailty intervention measures — Providing specialized guidance:
  * Physical Function and Fall History:
    * Prioritizing home safety for those with physical impairments.
    * Arranging rehab consultations when necessary.
  * Nutrition:
    * Assessing diets and offering education.
    * Pre-treatment nutritionist assessments.
    * Monitoring weight, intervening if >5-10% loss, or >10% loss.
  * Social Support:
    * Evaluating the needs of those without family support.
    * Referring to social services and introducing care resources.
  * Cognition:
    * Detecting cognitive issues, addressing reversible causes.
    * Assessing decision-making and medication self-administration.
    * Refer to specialists when needed.
  * Polypharmacy and Comorbidity:
    * Collecting medication data, ensuring adherence.
    * Noting chronic illnesses.
    * Collaborating with specialists or pharmacists for complex cases.
  * Psychological:
    * Providing weekly support for psychological concerns.
    * Refer to specialists for assessments and treatment options.
  Arms: Frail group

SUMMARY:
Gastric cancer ranks among the top ten leading causes of death in Taiwan. Radical surgery is the sole curative method for gastric cancer. However, our previous research has revealed that elderly gastric cancer patients undergoing radical surgery face a significantly elevated risk of postoperative complications. Even after gastric cancer resection, only 70% of patients receive adjuvant chemotherapy, with a particularly low likelihood among those aged ≥ 65 to undergo such treatment. With the increasing elderly population in our country, an increasing number of elderly gastric cancer patients must decide whether they can withstand radical surgery for gastric cancer and whether to undergo adjuvant chemotherapy. Therefore, increasing the rates of elderly gastric cancer patients undergoing radical surgery and adjuvant chemotherapy, as well as improving the success rate of chemotherapy, has become a critical issue.

Frailty has been a frequent topic in geriatric medicine in recent years. It involves assessing multifaceted aspects of physical functioning to determine an individual's frailty status, which can help predict the likelihood of severe side effects from medical interventions. International organizations like the American Cancer Society recommend frailty assessment for all elderly cancer patients before undergoing chemotherapy and corresponding interventions to address frailty. However, there is a lack of large-scale studies on frailty assessment and its practical clinical benefits in our population.

This study is a prospective, open-label, randomized clinical trial designed to investigate the impact of geriatric intervention on the tolerance of surgery/chemotherapy in patients diagnosed with gastric cancer. As part of the study protocol, all enrolled patients will undergo a comprehensive frailty assessment within a window of 7 days before initiating their first treatment, followed by tailored geriatric interventions.

The primary objective of this study is to assess and compare the effects of geriatric intervention on postoperative complications, chemotherapy tolerance, treatment-related toxicity, and overall quality of life among two distinct groups: frail and non-frail patients. Our research team aims to promote widespread frailty assessment and interventions with the following objectives:

1. Reduce the probability of postoperative complications among elderly gastric cancer patients receiving surgery.
2. Enhance the tolerance and success rate of adjuvant chemotherapy for gastric cancer.

These efforts ultimately aim to improve the survival prognosis of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged sixty-five or older with locally advanced (stage II and stage III) gastric cancer, preparing for curative gastric cancer surgery and scheduled to receive adjuvant chemotherapy within 4-8 weeks postoperatively, either as outpatients or inpatients.
* Patients must provide signed informed consent.
* Estimated survival of more than 3 months.
* Conscious and able to communicate verbally or in writing, and willing to cooperate with invasive procedures.

Exclusion Criteria:

* Patients with cognitive impairment or unable to cooperate with the interventional procedures as determined by the clinical physician.
* Patients receiving concurrent other anticancer treatments (radiation or surgery).
* Patients with multiple types of cancer requiring simultaneous treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing surgical complications between frail and non-frail patients using the Clavien-Dindo grading system. | After completion 3 months treatment.
Utilize CTCAE v5.0 to assess the grade and frequency of adverse events and treatment-related toxicity in frail and non-frail patient groups, and compare the differences between the two. | After completion 3 months treatment.

SECONDARY OUTCOMES:
Examine whether implementing appropriate frailty interventions can reduce the likelihood of adverse events, as assessed by the Clavien-Dindo grading system or CTCAE v5.0, occurring in frail groups three months after initiating treatment. | After completion 6 months treatment.
  The frail group will receive management and recommendations based on the specific impairment domain.
To compare overall survival between two distinct groups: frail and non-frail patients. | up to 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan